CLINICAL TRIAL: NCT01303627
Title: The Effects of Maintenance a Remifentanil Infusion on the Hemodynamic Variables and Recovery Quality
Brief Title: Safety of Remifentanil Infusion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, derya özkan, MD consultant, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DiskapiTRH
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Results first posted 2012-06-18 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-06

CONDITIONS: Urinary Tract Problem
Keywords: Remifentanil; Laryngeal mask airway removal; Hemodynamic changing; Infusion; Ureterorenoscopy
MeSH Terms: interventions — Remifentanil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ultiva,remifentanil,opioid,analgesic (Active Comparator): Remifentanil:1.5ng/ml remifentanil infusion maintained at the end of the surgery
  Interventions: Drug: remifentanil
- control (No Intervention): Control:Remifentanil stopped at the end of the surgery

INTERVENTIONS:
Drug: remifentanil — 1-4 ng/mL i.v. infusion during the surgery, maintenance dosage till LMA removal is 1.5 ng/mL.
  Arms: ultiva,remifentanil,opioid,analgesic

SUMMARY:
The effect of maintenance remifentanil infusion with target controlled infusion during laryngeal mask airway removal on hemodynamic parameters and emergence quality is going to be investigated.

DETAILED DESCRIPTION:
In all patients (control group and remifentanil group induction of anesthesia will be achieved with desflurane and remifentanil.Anesthesia will be maintained with remifentanil (1-4 ng/mL) by TCI target controlled infusion, and desflurane . Throughout the surgery hemodynamic parameters are going to be recorded. As soon as the surgery has been finished, in control group remifentanil infusion and desflurane inhalation is going to be stopped.In remifentanil group,desflurane inhalation is going to be stopped and remifentanil infusion will be maintained until the removal of LMA. During the emergence period the time of eye opening, hemodynamic parameters and emergence quality (score 1-2)are going to be recorded.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II status
* aged 18-60 years old
* presenting for ureterorenoscopy

Exclusion Criteria:

* history of hypertension
* asthma and chronic obstructive lung disease
* recent respiratory tract infections

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2011-02; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jülide Ergil, MD, Study Chair — Ministry of Health Dıskapi Yildirim Beyazit Training and Research Hospital, Anesthesiology 1.; Alp Alptekin, MD, Study Chair — Ministry of Health Diskapi Yildirim Beyazit Training and Research Hospital, Anesthesiology 1; Nihan Aktürk, MD, Study Chair — Ministry of Health Diskapi Yildirim Beyazit Training and Research Hospital , Anesthesiology 1; Haluk Gümüs, MD, Study Chair — Ministry of Health Diskapi Yildirim Beyazit Training and Research Hospital, Anesthesiology 1
Locations (1):
- Ministry of Health Diskapi Yildirim Beyazit Research and Training Hospital departement of 1. Anesthesiology, Ankara, Turkey (Türkiye)

REFERENCES:
- [Result] Nho JS, Lee SY, Kang JM, Kim MC, Choi YK, Shin OY, Kim DS, Kwon MI. Effects of maintaining a remifentanil infusion on the recovery profiles during emergence from anaesthesia and tracheal extubation. Br J Anaesth. 2009 Dec;103(6):817-21. doi: 10.1093/bja/aep307. Epub 2009 Oct 28. PMID 19864308

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ultiva,Remifentanil,Opioid,Analgesic | Control
Started | 21 | 21
Completed | 21 | 20 (One patient excluded from the study because of the failure while performing uretero-renoscopy)
Not Completed | 0 | 1
Not completed — the failure while performing URS | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ultiva,Remifentanil,Opioid,Analgesic | Control | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 20 | 41
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 41 (13) | 38 (12) | 39 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 8
  Male | 19 | 14 | 33
Region of Enrollment [Number; unit: participants]
  Turkey | 21 | 20 | 41

OUTCOME MEASURES:

1. Primary Outcome: Smooth cLMA Removal Condition (Score 1)
Description: cLMA removal was accepted as successful (score 1) if none of the complications coughing, teeth clenching, gross purposeful movements, breath holding, laryngospasm, and desatura- tion to SpO2\90% was observed. If any of these compli- cations was observed it was regarded as unsuccessful (score 2)
Time Frame: At the end of the surgery
Measure: Number; unit: percentage of participants
Groups:
- Remifentanil Group: remifentanil group (group R) TCI effect-site of remifentanil at 1.5 ng/ml was continued until cLMA removal
- Control Group: Remifentanil stopped at the and of the surgery
Arm/Group | Remifentanil Group | Control Group
Number analyzed (Participants) | 21 | 20
percentage of participants | 86 | 40
Statistical Analysis 1: Comparison: Remifentanil Group vs Control Group; The incidence of complications on removal of the cLMA has been reported 54 % in awake patients group A power analysis indicated that a minimum 16 patients in each group were required to demonstrate a difference that 50% reduction the complications (a power of 80% and α error 0.05); Test type: Superiority or Other; p < 0.05, Chi-squared — Statistical analyses were performed x2 test or Mann Whitney U test as approriate. A p value of <0.05 was considered statistically significant

ADVERSE EVENTS:
Time Frame: During the surgery
Description: serious and/or other [non-serious] adverse events were not collected/assessed.
Groups:
- Control Group: Remifentanil stopped at the end of the surgery
Arm/Group | Remifentanil Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The limitation of our study is age and ASA status of the included patients'. The relatively older or ASA status III,IV population may interfere the effect-site concentration TCI of remifentanil

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No